CLINICAL TRIAL: NCT00867711
Title: Pharmacogenetics of Pemetrexed and Carboplatin in Malignant Pleural Mesothelioma Patients
Brief Title: Molecular Predictors of Pemetrexed and Carboplatin Response in Malignant Pleural Mesothelioma (MPM) Patients
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: ONC/OSS-04/2008
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: MALIGNANT PLEURAL MESOTHELIOMA
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The paraffin-embedded tumor specimens of patients will be collected. The tumor RNA and DNA will be extracted and genotyping, gene expression and gene copy number analyses will be performed with validated PCR and array-CGH techniques.
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the present study is to investigate the molecular predictors of pemetrexed and carboplatin response in tumor samples of a series of MPM patients extracting the DNA and genotyping for the TSER polymorphism.

DETAILED DESCRIPTION:
Malignant pleural mesothelioma (MPM) is an aggressive tumor that usually has a poor prognosis. The combination of cisplatin and pemetrexed has recently become the standard of care in the first-line treatment of MPM. For patients who are unfit to receive a cisplatin-based chemotherapy, pemetrexed alone [7] or combined with carboplatin [8] has been proposed as an alternative treatment choice. The identification of molecular predictors of effective therapy is important for maximizing therapeutic efficacy and minimizing useless treatment in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* MPM diagnosis
* Availability of tumor tissue to perform analysis

Exclusion Criteria :

* Other primary diagnosis
* No archival tissue available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Malignant Pleural Mesothelioma patients treated with carboplatin and pemetrexed
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the expression and allelic variants of a panel of candidate genes involved in the resistance to drugs, the genome wide copy number changes in patients treated with drugs combination in the first line | one year

SECONDARY OUTCOMES:
Evaluate retrospectively the correlation between gene expression and polymorphisms in candidate genes and array-CGH data, immunohistochemistry data, and clinical data. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

REFERENCES:
- [Derived] Zucali PA, Giovannetti E, Destro A, Mencoboni M, Ceresoli GL, Gianoncelli L, Lorenzi E, De Vincenzo F, Simonelli M, Perrino M, Bruzzone A, Thunnissen E, Tunesi G, Giordano L, Roncalli M, Peters GJ, Santoro A. Thymidylate synthase and excision repair cross-complementing group-1 as predictors of responsiveness in mesothelioma patients treated with pemetrexed/carboplatin. Clin Cancer Res. 2011 Apr 15;17(8):2581-90. doi: 10.1158/1078-0432.CCR-10-2873. Epub 2011 Jan 24. PMID 21262916